CLINICAL TRIAL: NCT02553252
Title: Sudarshan Kriya Yoga (SKY) Versus Wait List Control (WLC) in Post Traumatic Stress Disorder: A Randomised Controlled Study
Brief Title: SKY Versus WLC in PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A pilot study is currently in progress.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Kamini Vasudev, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106851
Record Dates: First submitted 2015-09-05; First posted 2015-09-17 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Post Traumatic Stress Disorder
Keywords: post traumatic stress disorder (PTSD); Sudarshan Kriya Yoga (SKY)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sudarshan Kriya Yoga Trauma Relief Program (SKY) (Experimental): Participants will receive training in SKY soon after completing baseline assessments.
  Interventions: Other: Sudarshan Kriya Yoga Trauma Relief Program (SKY)
- wait list control (WLC) (No Intervention): Participants will receive training in SKY after 12 weeks have passed since the baseline assessment.

INTERVENTIONS:
Other: Sudarshan Kriya Yoga Trauma Relief Program (SKY) — Participants in the SKY group will undergo a 12-week training course in Sudarshan Kriya Yoga (SKY) conducted by certified instructors from the Art of Living Foundation.
  Arms: Sudarshan Kriya Yoga Trauma Relief Program (SKY)

SUMMARY:
Patients with post traumatic stress disorder (PTSD) will be randomized to a 12-week intervention of Sudarshan Kriya Yoga Trauma Relief Program (SKY) or a wait list control (WLC) to assess the effects of this intervention on symptoms of PTSD, depression, anxiety, quality of life, autonomic symptoms, and blood inflammatory markers.

DETAILED DESCRIPTION:
A single-center, single blind longitudinal randomized controlled naturalistic trial comparing a 12 week Sudarshan Kriya Yoga Trauma Relief Program (SKY) intervention to a wait list control (WLC) group.

Research participants will be men and women, 18-75 years of age, who have PTSD. The study will recruit from the general adult ambulatory mental health clinics as well as the geriatric mental health program in London.

Potential participants will be screened as per inclusion and exclusion criteria by trained research staff. These patients will already have clinically diagnosed PTSD by a psychiatrist and any other comorbid diagnoses would have already been confirmed. However, for research purposes a diagnosis of PTSD will be confirmed through a structured clinical interview specifically the MINI (Mini International neuropsychiatric Interview) and the Clinician-administered PTSD Scale for DSM5- past month version (CAPS5). CAPS5 will also be used to rule out exclusion criteria of severe depersonalization and derealization. The scales will be administered by a trained research staff and confirmed by a psychiatrist.

The MINI will also be used to assess for suicidality. If the total score on Questions C1 and C2 is more than 5 at any time during the study then this will be reported to the PI who will further assess the patient for safety and risk assessment.

If the participant is above the age of 65 years of age they will also be asked to complete a cognitive screening test (Mini Mental State Examination, MMSE) to ensure they are not suffering from any memory impairments.

Participants who meet the inclusion criteria will be randomized to either SKY or WLC with equal probability (1:1) using computer generated randomisation numbers. Concealment of randomisation to outcome assessors and investigators will be ensured by an independent staff member who will perform the randomisation using a third party web based provider. Computerised randomization will take place in the Geriatric Mental Health Program outpatient unit in London Health Sciences, London, Ontario. A telephone number will be available for study concerns/queries. Pre-randomized information will be stored using unique de-identifiers and downloaded on a secure database. It will not be possible to blind participants to intervention status hence the single-blind design.

SKY training involves attending a week-long (6 days) course that teaches the basic principles of SKY over 2.5-3 hour daily sessions. This will be followed by once weekly follow up sessions (90 min/wk) for 3 weeks and then bimonthly sessions (every 2 weeks) for the next 8 weeks. In addition, participants will be asked to practice SKY at home daily (25 min/day) throughout the duration of the study period and log practice frequency and any other noteworthy observations in a log sheet that will be provided to them (please see attached log sheet). Meals will be provided for 2 days during the initial SKY training course and nutritional snacks on the other 4 days.

Participants randomized to the control arm of the study will continue to receive their treatment as usual, including pharmacotherapy and/or psychotherapy. They will follow assessment and study procedures as listed below. Upon completing the initial 12 weeks of the study, participants in the WLC arm will also be offered the opportunity to learn SKY and attend follow up therapy sessions; that is, WLC participants will be offered the same intervention as the SKY group received in the first 12 weeks of the study. No study procedures will be applied or any other information collected during this period except for a final assessment that will take place at 24 weeks (see below).

ELIGIBILITY:
Inclusion Criteria:

1. Have an Axis 1 diagnosis of PTSD as per CAPS5 (Clinician Administered PTSD Scale for DSM 5- past month version) criteria.
2. If participants are using antidepressants, they must be at therapeutic doses for a minimum of four weeks prior to commencing the study. Patients who are not willing to take any medications will also be eligible for the study
3. Sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 60 minutes.
4. Willing and able to attend 6 initial SKY training sessions and 75% of follow up sessions
5. Not pregnant and willing to remain not pregnant for the duration of the study

Exclusion Criteria:

1. They are currently participating in other similar studies.
2. If the patient scores severe or extreme on Depersonalization (item 29) or Derealization (item 30) items of CAPS5.
3. Other significant mental health diagnosis including substance dependence, Neurocognitive disorder, Obsessive Compulsive Disorder, Panic Disorder, Bipolar disorder and/or Personality disorder (confirmed by Psychiatrist and MINI)
4. High risk of suicide as elicited by clinical interview (MINI).
5. Psychotic episodes within the past 12 months.
6. Traumatic Brain Injury (TBI) as defined by loss of consciousness for more than 20 minutes and/or Glasgow Coma Scale score less than or equal to 12. (The researcher will use self-reported histories to screen for traumatic brain injury and if necessary confirmed by medical records.
7. Currently practicing any type of formal meditation, mindfulness or breathing techniques regularly.
8. Serious cardiovascular disease in the past 12 months (i.e. myocardial infarction, stroke, TIA, uncontrolled hypertension), or a past history of neurological disease (including Parkinson's Disease), seizures, or diabetic neuropathy
9. Major surgery within 6 weeks prior to commencement of the intervention, or a scheduled major surgery during the intervention period. (This is due to the physical rigor of the breathing techniques).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Reduction in PTSD symptoms as assessed by the clinician administered PCL-5 (Post Traumatic Stress Disorder Check List). | Change from baseline to: 4 weeks, 8 weeks, 12 weeks, and 24 weeks
  The clinician administered PCL-5 (Post Traumatic Stress Disorder Check List). willl be used to assess a change in PTSD symptoms from baseline to weeks 4, 8, 12, and 24.

SECONDARY OUTCOMES:
Reduction in depression symptoms as assessed by the clinician administered HAM-D 17 (Hamilton Depression Score). | Change from baseline to: 4 weeks, 8 weeks, 12 weeks, and 24 weeks
  A clinican administered depression severity assessment scale HAM-D 17 will be used to assess the change in depression symptoms from baseline to weeks 4, 8, 12, and 24.
Reduction in anxiety symptoms as assessed by the HAM-A (Hamilton Anxiety Scale). | Change from baseline to: 4 weeks, 8 weeks, 12 weeks, and 24 weeks
  A clinician administered Hamilton Anxiety Scale (HAM-A) will be used to assess a change in anxiety symptoms from baseline to weeks 4, 8, 12, and 24.
Improvement in autonomic parameters including heart rate variability and heart rate as assessed by a Bluetooth enabled Polar H7 Heart Rate Sensor. | Change from baseline to: 12 weeks, and 24 weeks.
  Heart rate and heart rate variability will be measured to assess a change from baseline to weeks 12 and 24 in autonomic parameters.
Improvement in blood inflammatory markers as measured by enzyme-linked immunosorbent assay. | Change from baseline to: 12 weeks, and 24 weeks.
  A blood sample will be taken to run an enzyme-linked immunosorbent assay (ELISA) to assess levels of the following inflammatory markers: C-Reactive Protein (CRP), Interleukin-6 (IL-6), malondialdehyde (MDA) and total antioxidant capacity (including glutathione). This will be done at baseline, week 12, and week 24 to assess a change in blood inflammatory markers.
Reduction in depression symptoms using self-rated BDI 21 (Beck's Depression Inventory). | Change from baseline to: 4 weeks, 8 weeks, 12 weeks, and 24 weeks
  A self-administered depression severity assessment scale BDI 21 will be used to assess the change in depression symptoms from baseline to weeks 4, 8, 12, and 24.
Change in quality of life as assessed by the WHOQOL-Bref (World Health Organization Quality of Life Scale). | Change from baseline to: 4 weeks, 8 weeks, 12 weeks, and 24 weeks
  The WHOQOL-Bref will be used to assess any changes in quality of life from baseline to weeks 4, 8, 12, and 24.
Improvement in blood pressure as assessed by manually using a standard plethysmograph. | Change from baseline to: 12 weeks, and 24 weeks.
  A research assistant will manually obtain 3 blood pressures at each blood pressure assessment. The mean will be calculate from the three measurements and used to assess a change in blood pressure from baseline to weeks 12 and weeks 24.
Improvement in the mean respiratory rate as measured manually. | Change from baseline to: 12 weeks, and 24 weeks.
  The mean respiratory rate will be calculated from three readings taken at each of the respiratory rate assessments (baseline, week 12, and week 24). The research assistant will record the number of breaths per minute, each breath consisting of an inhalation and exhalation.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, LHSC, London, Ontario, Canada